CLINICAL TRIAL: NCT01634334
Title: Innovation for Smoke-Free Homes: Real-Time Feedback
Brief Title: Improving Household Air Quality in Homes With Children
Acronym: ProjFreshAir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Melbourne Hovell, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL103684 (NIH)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Lung Diseases; Asthma
Keywords: Secondhand smoke
MeSH Terms: conditions — Lung Diseases; Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real-time Intervention (Experimental)
  Interventions: Behavioral: Real-Time Intervention
- Usual Education (Active Comparator): Participants will receive usual education about secondhand and thirdhand smoke.
  Interventions: Behavioral: Usual Education

INTERVENTIONS:
Behavioral: Real-Time Intervention — Lights and Sound Brief Coaching
  Arms: Real-time Intervention
Behavioral: Usual Education — Participants will receive usual education about secondhand smoke and thirdhand smoke.
  Arms: Usual Education

SUMMARY:
The purpose of this study is to determine if real-time feedback (lights/sounds) from small smoke particle monitors and brief coaching will encourage parents to reduce young children's secondhand tobacco smoke exposure in their home.

DETAILED DESCRIPTION:
The purpose of this efficacy study is to test whether children's home secondhand tobacco smoke exposure (measured by cotinine & nicotine assays, fine particulates and reports of smoking in the home and/or home smoking bans) can be reduced by using custom particle monitors to provide real-time feedback to household residents plus brief advice/praise.

ELIGIBILITY:
Inclusion Criteria:

* Families with at least one parent or guardian (18 years of age or older),
* Household resident who smokes tobacco,
* Child under fourteen years old exposed to tobacco smoking in the home
* Plans to live in San Diego County for at least three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Secondhand Smoke Reduction | Measured from baseline upto 5 months
  Parental report and child urine cotinine.

SECONDARY OUTCOMES:
Home Smoking Ban | Measured from baseline upto 5 months.
  Parental report of home smoking ban and environmental data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne F Hovell, PhD, MPH, Principal Investigator — SDSU - Center for Behavioral Epidemiology and Community Health
Locations (1):
- SDSU - Center for Behavioral Epidemiology and Community Health, San Diego, California, United States

REFERENCES:
- [Derived] Hovell MF, Bellettiere J, Liles S, Nguyen B, Berardi V, Johnson C, Matt GE, Malone J, Boman-Davis MC, Quintana PJE, Obayashi S, Chatfield D, Robinson R, Blumberg EJ, Ongkeko WM, Klepeis NE, Hughes SC; Fresh Air Research Group. Randomised controlled trial of real-time feedback and brief coaching to reduce indoor smoking. Tob Control. 2020 Mar;29(2):183-190. doi: 10.1136/tobaccocontrol-2018-054717. Epub 2019 Feb 15. PMID 30770436
- [Derived] Hughes SC, Bellettiere J, Nguyen B, Liles S, Klepeis NE, Quintana PJE, Berardi V, Obayashi S, Bradley S, Hofstetter CR, Hovell MF. Randomized Trial to Reduce Air Particle Levels in Homes of Smokers and Children. Am J Prev Med. 2018 Mar;54(3):359-367. doi: 10.1016/j.amepre.2017.10.017. Epub 2018 Jan 2. PMID 29305069